CLINICAL TRIAL: NCT04441424
Title: The Therapeutic Potential of Convalescent Plasma Therapy on Treating Critically-ill COVID-19 Patients Residing in Respiratory Care Units in Hospitals in Baghdad, Iraq
Brief Title: Convalescent Plasma Therapy on Critically-ill Novel Coronavirus (COVID-19) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alkarkh Health Directorate-Baghdad (Other Government)
Responsible Party: Principal Investigator, Ahmed Sahib Abdulamir, Professor in Virology and infectious diseases, Alkarkh Health Directorate-Baghdad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CPT-COVID-19
Record Dates: First submitted 2020-06-12; First posted 2020-06-22 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: IMMUNOTHERAPY
MeSH Terms: interventions — Hydroxychloroquine; Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Convalescent plasma group (Experimental): 21 critically-ill COVID-19 patients were given convalescent plasma: 400 ml of convalescent plasma from COVID-19 recovered subjects. The plasma infusion lasts for one hour.
  Interventions: Biological: Convalescent plasma; Drug: Hydroxychloroquin with Azithromycin
- Control group (Other): This group is 28 critically-ill COVID-19 patients who are at the same disease stage to those of experimental group that were treated with conventional therapy without taking convalescent plasma.
  The conventional therapy: 400 mg once PO Hydroxychloroquine/day with 250mg once PO Azithromycin.
  Interventions: Drug: Hydroxychloroquin with Azithromycin

INTERVENTIONS:
Biological: Convalescent plasma — 400 ml of convalescent plasma (plasma taken 2 weeks from the recovered COVID-19 patients) and was transfused over 1-2 hours to the recipients by blood donation set.
  Arms: Convalescent plasma group
Drug: Hydroxychloroquin with Azithromycin — The control group of COVID-19 patients were given the conventional therapy approved in Iraq for COVID-19, namely Hydroxychloroquine 400mg PO twice per day for 5 days and Azithromycin once PO 500 mg per day for 5 days.

SUMMARY:
Out of 49 early-stage critically-ill COVID-19 patients, 21 patients are the experimental group who take convalescent plasma compared to 28 patients receive only conventional therapy without taking Convalescent plasma. Recovery or death, length of stay in hospital, and improvement in the clinical course of the disease are monitored in relation to monitoring through severe acute respiratory syndrome Coronavirus 2 (SARS-CoV-2) RNA detection via poly chain reaction (PCR), and SARS-CoV-2 immunoglobulin G (IgG) and immunoglobulin M (IgM) serological monitoring.

DETAILED DESCRIPTION:
Objectives: The current COVID-19 pandemic needs unconventional therapies to tackle the resulted high morbidity and mortality. Convalescent plasma is one of the therapeutic approaches that might be of benefit. Methods: Forty nine early-stage critically-ill COVID-19 patients residing in respiratory care units (RCU) of three hospitals in Baghdad, Iraq were included, 21 received convalescent plasma while 28 did not receive, namely control group. Recovery or death, length of stay in hospital, and improvement in the clinical course of the disease were monitored clinically along with laboratory monitoring through SARS-CoV-2 RNA detection via PCR, and SARS-CoV-2 IgG and IgM serological monitoring.

ELIGIBILITY:
Inclusion Criteria:

* 49 critically-ill COVID-19 patients are included.
* All of the patients were with pneumonia and residing in RCU
* Age ≥ 18 y
* With dyspnea and oxygen saturation less than 90% in resting state.
* At their first 3 days in RCU either receiving O2 therapy, c-pap, or on ventilators.
* All of the patients were residing in infectious diseases wards before being transferred to RCU.

Exclusion Criteria:

* The exclusion criteria of the COVID-19 patients were:

  * Previous allergic history to plasma or its ingredients such as sodium citrate.
  * Cases with serious general conditions, such as severe organ dysfunction, that are not suitable for transfusion.
  * Very late stage of the acute respiratory distress (ARDS) where Convalescent plasma (CP) has proved to be of low therapeutic benefit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2020-04-03 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Death versus survival of treated patients | Up to 8 weeks
  evaluate the role of convalescent plasma in saving life of treated patients by measuring the final outcome whether treated patients survived or died

SECONDARY OUTCOMES:
The length of stay in hospitals | Up to 8 weeks
  this outcome is about measuring the length of stay (in days) of treated patients with convalescent plasma versus tose who were treated with conventional therapies

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed S Abdulamir, PhD, Principal Investigator — Alkarkh health directorate
Locations (1):
- Akarkh Healt hdirectorate, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Iannizzi C, Chai KL, Piechotta V, Valk SJ, Kimber C, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Jindal A, Cryns N, Estcourt LJ, Kreuzberger N, Skoetz N. Convalescent plasma for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2023 May 10;5(5):CD013600. doi: 10.1002/14651858.CD013600.pub6. PMID 37162745
- [Derived] Iannizzi C, Chai KL, Piechotta V, Valk SJ, Kimber C, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Jindal A, Cryns N, Estcourt LJ, Kreuzberger N, Skoetz N. Convalescent plasma for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2023 Feb 1;2(2):CD013600. doi: 10.1002/14651858.CD013600.pub5. PMID 36734509
- [Derived] Piechotta V, Iannizzi C, Chai KL, Valk SJ, Kimber C, Dorando E, Monsef I, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Estcourt LJ, Skoetz N. Convalescent plasma or hyperimmune immunoglobulin for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2021 May 20;5(5):CD013600. doi: 10.1002/14651858.CD013600.pub4. PMID 34013969
- [Derived] Chai KL, Valk SJ, Piechotta V, Kimber C, Monsef I, Doree C, Wood EM, Lamikanra AA, Roberts DJ, McQuilten Z, So-Osman C, Estcourt LJ, Skoetz N. Convalescent plasma or hyperimmune immunoglobulin for people with COVID-19: a living systematic review. Cochrane Database Syst Rev. 2020 Oct 12;10:CD013600. doi: 10.1002/14651858.CD013600.pub3. PMID 33044747

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-01): https://cdn.clinicaltrials.gov/large-docs/24/NCT04441424/Prot_SAP_000.pdf